CLINICAL TRIAL: NCT03850587
Title: A Multi-center, Double-blinded, Randomized, Active-controlled, Parallel Design, phaseII Study to Investigate the Efficacy and Safety of YYC301 in Subject With Knee Osteoarthritis.
Brief Title: Clinical Trial of YYC301 for Treatment of Osteoarthritis of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yooyoung Pharmaceutical Co., Ltd. (Industry)
Collaborators: CliPS Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YYPCT_YYC301_P2
Record Dates: First submitted 2019-02-20; First posted 2019-02-22 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Celecoxib; Tramadol

STUDY DESIGN:
Intervention Model Description: The purpose of this study is to investigate the efficacy and safety after administration of YYC301(Experimental) or Celecoxib(Comparator) in subjects with knee osteoarthritis in a state of uncontrolled pain who took Celecoxib(Cox-2 inhibitor).
Who Masked: Participant, Investigator
Masking Description: double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- YYC301-1 & Celocoxib placebo (Experimental): YYC301-1 one capsule and Concomitant Drug Celocoxib placebo.
  *YYC301-1 is a capsule. It is composed of Celocoxib 200mg and Tramadol 37.5mg complex).
  Interventions: Drug: Tramadol 37.5Mg+ Celecoxib 200mg
- YYC301-2 & Celocoxib placebo (Experimental): YYC301-2 one capsule and Concomitant Drug Celocoxib placebo.
  *YYC301-2 is a capsule. It is composed of Celocoxib 200mg and Tramadol 75mg complex)
  Interventions: Drug: Tramadol 75mg+ Celecoxib 200mg
- YYC301-3 & Celocoxib placebo (Experimental): YYC301-3 one capsule and Concomitant Drug Celocoxib placebo.
  *YYC301-3 is a capsule. It is composed of Celocoxib 200mg and Tramadol 150mg complex)
  Interventions: Drug: Tramadol 150mg+ Celecoxib 200mg
- YYC301 placebo & Celecoxib (Active Comparator): Concomitant Drugs with Celecoxib 200mg and YYC301 one capsule.
  Interventions: Drug: Celecoxib 200mg

INTERVENTIONS:
Drug: Celecoxib 200mg — comparator medication
  Arms: YYC301 placebo & Celecoxib
Drug: Tramadol 37.5Mg+ Celecoxib 200mg — experimental medication
  Other Names: yyc301-1
  Arms: YYC301-1 & Celocoxib placebo
Drug: Tramadol 75mg+ Celecoxib 200mg — experimental medication
  Other Names: yyc301-2
  Arms: YYC301-2 & Celocoxib placebo
Drug: Tramadol 150mg+ Celecoxib 200mg — experimental medication
  Other Names: yyc301-3
  Arms: YYC301-3 & Celocoxib placebo

SUMMARY:
A Multi-center, Double-blinded, Randomized, Active-controlled, Parallel Design, phaseII Study to Investigate the Efficacy and Safety of YYC301 in Subject With Knee Osteoarthritis

ELIGIBILITY:
Inclusion Criteria:

* Men/Women aged over 20
* Subjects who are diagnosed with one- or both-sided knee osteoarthritis according to the standards of clinical diagnosis from American College of Rheumatology(ACR)have knee osteoarthritis pain and meet over three of the following conditions.

  1. Older than 50
  2. Morning stiffness for less than 30 minutes
  3. Crepitus on active motion
  4. Bony tenderness
  5. Bony enlargement
  6. Not have heat-generating site
* Subjects who are diagnosed with degenerative osteoarthritis and have its pain at least for over 3 months before the screening visit.
* Subjects who are uncontrolled with pain after administration of Celecoxib at least for over 2 weeks before the randomization and have more than 40mm out of 100mm VAS at randomization.
* Subjects who voluntarily agree to participate in this clinical trial in writing.

Exclusion Criteria:

* Subjects with rheumatoid arthritis or inflammatory, infectiousand metabolic arthritis.
* Subjects with ochronosis, hemochromatosis, secondary knee osteoarthritis by systemic disease.
* Subjects who have severe pain such as Sudek's atrophy, Paget's disease and spinal disc herniation.
* Subjects with poly-articular affected by severe pain of knee osteoarthritis.
* Subjects who take psychtrophic medicine and narcotic analgesics for over 3 months that might affect on pain sensory system.
* Subjects who had Tramadol but there was no improvement in pain.
* Subjects who got the follwing treatment and medicine before the screening;

  1. Subjects who had surgery on knee ligaments within a year, cartilage transplant and scarf osteotomy.
  2. Subjects who had arthroscopy within 6 months.
  3. Subjects with intra-articular knee joint steroid injection within 3 months.
  4. Subjects with HA injection in knee joint within 2 months.
  5. Subjects with systemic steroid injection within a month(but inhaled steroids)
  6. Subjects with knee replacement surgery.
* Subjects who hot the following treatment and medicine before the randomization;

  1. Subjects who had Celecoxib, acetaminophen or steroidal/non-steroidal anti-inflammatory drugs except low dose aspirin(before 300mg/day) But, acetaminophen and low dose aspirin (before 300mg/day) are prohibited within 24 hours)
  2. Nutritional supplements, physical therapy and Korean herbal medicine for knee osteoarthritis and it pain within 2 weeks.
* Subjects who have to take anticoagulant drugs such as warfarin and coumarin during this clinical trial.
* Subjects who took MAO inhibitors within 14 days before the screening or needed to take these drugs during this clinical trials.
* Subjects with drug and opioid hypersensitivity and who have history.
* Subjects with sulfanilamide allergy and who have history.
* Subjects with asthmma, acute rhinitis, nasal polyp, angioedema, urticaria, allergic reaction to aspirin or any oher NSAIDs(incluing COX-2 inhibitors)
* Subjects with significant investigations - Hyperkalemia(Exceeded 5.5mmol/L)
* Subjects with severe liver dysfunction (ALT or AST of more than 3.0 times the upper limit of ULN and 1.5 tmines the upper limit of ULN)
* Subjects with severe renal impairment (Serum Creatine > 3x ULN).
* Subjects with active peptic ulcer and gastrointestinal bleeding.
* Severe blood disease (Agranulocytosis, aplastic anemia, hemolytic anemia, Thrombocytopenia, etc.).
* Subjects with Crohn's disease or inflammatory bowel disease such as ulcerative clitis.
* Subjects with congestive heart failure(NYHA 2-4)
* Subjects with severe ischaemic heart disease, peripheral artery disease and/or cerebrovascular disease.
* Subjects with genetic problesa such as galactose intolerance), lapp lactase deficiency or glucose-galactose malabsorption).
* Subjects with acute alcohol intoxification.
* Subjects who are addicted with took central nervous system drugs such as painkillers, sleeping pills, anti-anxiety medications, etc.
* Subjects with severe bronchopulmonary dysplasia.
* Subjects with head injury history of brain structure lesions which may be in danger of mental confusion.
* Subjects with epilepsy who are treated properly.
* Subjects who use Tramadol to cure for narcotic withdrawal.
* Subjects who took other clinical drugs more than once within 30 days before the clinical trial.
* Subjects suspected to be pregnant who don't agree with the clinical method which is permitted medically during clinical trial(Method of hormone contraception, IUD(Intrauterine device) or IUS(Intrauterine system)), tubal ligation, bilateral tubal ligation(condom, Diaphragm, etc).
* Pregnant woman and breastfeeding woman.
* Subjects who can increase risk due to clinical test and administraion of drugs or have severe grade / chronic medical, mental condition or abnormal laboratory result that may interfere with the analysis of thest results.
* Any other ineligible condition at the direction of investigator that would be ineligible to participate the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2020-05-12 (Actual); Study Completion 2020-09-07 (Actual)

PRIMARY OUTCOMES:
100mm Pain VAS | at 1,4,8,12 weeks after randomization after administration of YYC301(Experimental drug).
  Subjects who have severe pain at one-or both sided knee osteoarthritis directly assess the degree of pain (within 24 hours) with a straight line which has 0mm to 100mm. 0 mm means 'doesn't have pain' and 100 mm means 'maximum pain who can imagine'.In order to investigate the degree of subject's pain change from administration of YYC301(Experimental drug).
KOOS(Knee Injury and Osteoarthritis Outcome Score) | at 4,8,12 weeks after randomization after administration of YYC301(Experimental drug).
  KOOS survey is consisted of total 42 questions at 5 groups. 7 questions about symptoms, 9 questions about pain, 17 questions about Function in daily,5 questions about function in sport and recreation(sport/Rec), 4 questions about the knee related quality of life(QoL). Subjects who are participated in this clinical trial, they directly assess these survey with 5 point Likert scale(0~4, 0 means 'nothing' and 4 means 'most severe') and KOOS results are converted to WOMAC score.
Patient Global Assessment(PGA) | at 4,8,12 weeks after randomization after administration of YYC301(Experimental drug).
  Subjects who have been admistrated YYC301 have to directly perform the patient global assessment with 5 point Likert Scale. It has 0 to 5 scales. 0 means 'very poor' and 5 means' very good' In order to investigate the Patient Global point assessment at specific weeks.
Total dosage and dosage rate of rescue treatment. | at screening time(visit 1; 2 weeks before next visit 2), randomization(visit 2), 4, 8 weeks after randomization.
  Subjects who administration of YYC301(Experimental drug) are investigated total dosage and dosage rate of rescue treatment.

CONTACTS AND LOCATIONS:
Locations (10):
- South Korea (10):
  - Dong-A University Hospital., Busan
  - Bundang Seoul University Hospital, Seoul
  - Gachon University Gil Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - KyungHee University Medical Center, Seoul
  - Soonchungyand University Hospital, Seoul
  - The Catholic University of Korea, Seoul ST. Mary's Hospital., Seoul